CLINICAL TRIAL: NCT05617794
Title: Effect of Diffusion Optics Technology (DOT) Spectacle Lenses on Choroidal Thickness and Choroidal Vascularity Index in Emmetropes
Brief Title: Effect of Diffusion Optics Technology (DOT) Spectacle Lenses on Choroidal Thickness
Acronym: ASH-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SightGlass Vision, Inc. (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CPRO-2207-001
Record Dates: First submitted 2022-11-01; First posted 2022-11-15 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Myopia; Myopia Progression; Juvenile Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Treatment 1 - Diffusion Optics Technology (DOT) Pattern (Experimental)
  Interventions: Device: Diffusion Optics Technology (DOT) Pattern Spectacle Lens
- Treatment 2 - Control Spectacles (Active Comparator)
  Interventions: Device: Control Spectacle Lens

INTERVENTIONS:
Device: Diffusion Optics Technology (DOT) Pattern Spectacle Lens — DOT Pattern Spectacle Lens
  Arms: Treatment 1 - Diffusion Optics Technology (DOT) Pattern
Device: Control Spectacle Lens — Control Spectacles
  Arms: Treatment 2 - Control Spectacles

SUMMARY:
The objective of the study is to measure the effect of Diffusion Optics Technology (DOT) spectacle lenses on the choroidal thickness and choroidal vascularity index compared to control lenses.

ELIGIBILITY:
Inclusion Criteria:

* Are 8-14 years of age;
* Are able to read (or be read to), understand and sign the assent document;
* Are accompanied by a parent or legal guardian who is able to read, understand and sign the parental information and permission document;
* Are emmetropic by non-cycloplegic auto-refraction, which means both refractive meridians should be within +1.00D and -1.00D inclusively;
* Are willing and able to follow instructions.

Exclusion Criteria:

* Are participating in any concurrent interventional clinical or research study;
* Have a history of myopia control treatment in the past year;
* Have amblyopia in either eye or known to have any other binocular vision disorder, such as accommodative insufficiency;
* Have any known active ocular disease and/or infection;
* Have a systemic condition that in the opinion of the investigator may affect a study outcome variable. Examples include diabetes mellitus, hyperthyroidism;
* Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable. Examples include Atropine eye drops;
* Have undergone strabismus surgery, refractive error surgery or intraocular surgery;
* Are a child of a member of the study team.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Choroidal Thickness | 30 minutes and 60 minutes
  Change from Baseline, 30 minutes and 60 minutes
Retinal and Choroidal Thickness | 30 minutes and 60 minutes
  Change from Baseline, 30 minutes and 60 minutes

SECONDARY OUTCOMES:
Software Method Comparison | 30 minutes and 60 minutes
  Comparison of measurements using different software methods; manual, semiautomated and automated software

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Ocular Research and Education, Waterloo, Ontario, Canada